CLINICAL TRIAL: NCT07361159
Title: Health and Wellness Coaching to Improve Thoracic Transplant Caregiver Self-Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-009890
Record Dates: First submitted 2025-12-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Wellbeing
Keywords: Health and Wellness Coaching; Thoracic Transplant; Caregivers; Caregiver Burden; Caregiver Self-efficacy
MeSH Terms: conditions — Caregiver Burden | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health and Wellness Coaching (Experimental): All caregiver participants will be in arm 1 and receive the health and wellness coaching intervention.
  Interventions: Behavioral: Health and Wellness Coaching

INTERVENTIONS:
Behavioral: Health and Wellness Coaching — Participants will receive health and wellness coaching. Coaching sessions will occur via telephone with a National Board-Certified Health and Wellness Coach (NBC-HWC). Sessions will be motivational interview based and will be up to 30 minutes in length. Participants can receive up to 8 coaching sessions within 10 weeks.
  Other Names: Health Coaching; Wellness Coaching

SUMMARY:
This is a pilot study examining the effects of telephonic health and wellness coaching on self-efficacy and caregiving burden for caregivers of patients awaiting heart or lung transplant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Primary caregivers of patients listed (active, deferred, or temporarily inactive) for lung, heart/lung, or heart transplantation at Mayo Clinic in Rochester

Exclusion Criteria:

* Individuals younger than 18 years old
* Individuals who are non-English speaking, non-verbal, or extremely hard of hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden Scale (CBS) | Completed at baseline and at study completion; 10 weeks after enrollment
  The CBS is a 21-item questionnaire where caregivers rate responses based on perceived level of burden on a 0-4 Likert scale. Scores are summed with higher scores indicating greater caregiver burden.
  No or minimal burden: 0 to 20 Mild to moderate burden: 21 to 40 Moderate to severe burden: 41-60 Severe burden: 61 to 88
Caregiver Self-Efficacy Scale | Completed at baseline and at study completion; 10 weeks after enrollment
  The Caregiver Self-Efficacy scale is a an 8-item questionnaire where caregivers rate their level of confidence on their ability to keep up with their own activities and caregiving situations using a 0-10 scale with 10 being totally confident. Total self-efficacy score is the mean of the eight items with higher scores indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No